CLINICAL TRIAL: NCT01197248
Title: Randomized Controlled Trial of Cystocele Plication Risks ("CPR Trial"): A Pilot Study
Acronym: CPR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Danny Lovatsis, Dr., Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPR Trial
Record Dates: First submitted 2010-08-17; First posted 2010-09-09 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Voiding Dysfunction
Keywords: cystocele; voiding; dysfunction
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystocele Plication (Active Comparator): Placement of sutures over the pubocervical fascia during cystocele repair.
  Interventions: Procedure: Cystocele plication
- No Plication (Experimental): Avoid sutures over pubocervical fascia during cystocele repair
  Interventions: Procedure: No Plication

INTERVENTIONS:
Procedure: Cystocele plication — placement of sutures over the pubocervical fascia during the cystocele repair
  Other Names: Cystocele reduction
  Arms: Cystocele Plication
Procedure: No Plication — Avoid sutures over pubocervical fascia during cystocele plication
  Other Names: No plicating sutures
  Arms: No Plication

SUMMARY:
Up to 50% of patients undergoing pelvic floor repair experience short-term postoperative voiding dysfunction, increasing the length of hospitalization, cost and anxiety among patients.

The mechanism behind this problem is the sutures placed in the pubocervical fascia during the cystocele repair. The cited benefit of bladder plication is greater cure of cystocele. The existence of pubocervical fascia and the need for placement of plicating sutures over the bladder have been questioned.

The objective of this study is to determine if avoiding cystocele plication in women undergoing surgery for cystocele decreases the need of catheterization beyond post operative day #2.

We will conduct a RCT of patients undergoing transvaginal repair of midline cystocele at the Mount Sinai Hospital. Patients will be randomized to receiving plicating sutures versus no plication. This procedure may be conducted with or without concomitant correction of other sites of prolapse. However, they will not have any procedures for correction of stress incontinence.

This study will be powered to detect a reduction in voiding dysfunction from 50% to 25% of patients. Using a χ2 distribution, and an alpha error of 0.05, the required sample size is 58 patients per group.

DETAILED DESCRIPTION:
Vaginal prolapse is a common problem in women. Approximately 11% of women undergo pelvic reconstructive surgery for either pelvic organ prolapse and/or urinary incontinence[1]. Several surgical techniques for correction of prolapse have evolved and have been scientifically evaluated. However, many basic surgical gynecological principles and techniques have been passed on over generations without any scientific evaluation. The technique of transvaginal repair of cystocele due to an anterior midline defect has traditionally included four steps: 1. mobilization of the defect (i.e. separation of vagina from bladder); 2. reduction of the defect (i.e. placement of plicating sutures into the pubocervical fascia); 3. trimming of redundant vaginal tissues; and 4. reapproximating the vaginal mucosa[2, 3]. Although each surgeon may modify any of these steps (ex. Depth of dissection, location and number of sutures), the principles are consistent. The existence of pubocervical fascia and the need for placement of plicating sutures over the bladder have been questioned, and some vaginal surgeons omit this step[4-6]. The cited benefit of bladder plication is greater cure of cystocele. Some of the potential risks of plication include ureteric obstruction, if the sutures are near the ureteric orifice, and voiding dysfunction if the sutures are near the urethrovesical junction[3, 7]. A chart review of patients at the Mount Sinai Hospital, who underwent typical pelvic floor repair, including transvaginal cystocele repair and mid-urethral sling, has shown that approximately 50% of patients experience short-term postoperative voiding dysfunction (non-published data), increasing the length of hospitalization, cost and anxiety among patients.

This pilot trial will assess the short-term risks of cystocele plication, and will assess trial feasibility. Ideally a larger subsequent trial will assess the cure of cystocele one year after surgery. To the best of my knowledge, this is the first study to assess the short-term post-operative outcomes in women who undergo this procedure.

3- Research Question In women with cystocele due to an anterior midline defect, does cystocele plication (independent variable) result in more or less patients requiring catheterization beyond postoperative day 2 (dependent variable) compared to no plication?

Hypothesis The hypothesis is that there may be more short-term voiding dysfunction and ureteric obstruction following cystocele repair with plication than following cystocele repair without plication.

4- Population of Interest and Sampling Methods Inclusion criteria: Patients between 18 and 75 years, who will undergo surgery at the Mount Sinai Hospital that includes cystocele repair, will be eligible.

Exclusion criteria: Patients will be excluded if the surgeon places anterior vaginal mesh or a mid-urethral sling, and/or if they had prior surgery for anterior vaginal wall prolapse and/or stress urinary incontinence.

Recruitment strategy: The patients will be recruited at the Mount Sinai Hospital Urogynecology Department. Approximately 4 to 6 eligible patients are seen per week and it is estimated that at least one patient will be recruited per week. The study will be completed in approximately two years. This will be a single centre study conducted at the Mount Sinai Hospital, Toronto, Canada.

5- Manoeuvre Study Design This study is a double blind, randomized controlled trial of patients undergoing transvaginal repair of midline cystocele, with or without concomitant correction of prolapse in other vaginal compartments, but without correction of stress incontinence. All the patients will provide written informed consent for participation. At baseline, all participants will undergo a standardized evaluation, which will include an urogynecologic history, pelvic organ prolapse quantification examination, and urodynamic evaluation. The urodynamic evaluation will include measurement of post-void residual urine volume by catheter and/or ultrasound bladder scan, uroflowmetry, a filling cystometrogram and urethral pressure profilometry.

Patients will be randomized intraoperatively using computer-based randomization. At the time of the surgical step of bladder plication, the computer program will be used, and will indicate whether sutures will be placed or omitted. Trimming of redundant vaginal mucosa will be performed before randomization to avoid any bias resulting from the amount of mucosa removed.

Standardized surgical technique

* Midline vaginal mucosal incision
* Sharp surgical dissection between vagina and pubocervical fascia.
* Completion of prolapse repair of vault, rectocele, uterine prolapse.
* Manual reduction of prolapse and trimming of redundant vaginal mucosa.
* Open envelope to determine group of allocation.
* If randomization to plication, place midline interrupted sutures of 0 or 2-0 polyglycolic acid sutures.
* Administer indigo carmine 5 ml IV.
* Cystoscopy with 70º telescopes.
* Close vaginal mucosa with running interlocking 0 or 2-0 polyglycolic sutures.

Protocol On postoperative day 1, patients will have the Foley catheter removed and measurement of post-void residual urine volume will be done (either by in and out catheterization, suprapubic ultrasound or via a Bonnano suprapubic catheter). Catheterization will be continued until residual volumes are less than 200 ml twice in a row. Registered nurses who will be masked to the treatment assignment will perform the post-operative assessment and examination.

6- Outcomes Primary Outcome Measures The primary outcome variable will be the requirement for catheterization beyond postoperative day 2. This has been chosen as the primary outcome since this would delay the usual hospital discharge on postoperative day 2, thus presenting a practical problem for patients (important based in our patients value and expectative after pelvic organ prolapse surgery), physicians, and hospitals (cost).

Other Outcome Measures A secondary outcome will be intraoperative ureteric obstruction. All patients, regardless of study arm, will undergo intraoperative cystoscopy following intravenous administration of indigo carmine in order to identify this complication. If this complication does occur the suspected plicating suture(s) will removed, replaced more centrally, and cystoscopy repeated to ensure ureteric permeability.

Analysis Sample Size A chart review of patients at the Mount Sinai Hospital, who underwent typical pelvic floor repair, including transvaginal cystocele repair and mid-urethral sling, has shown that approximately 50% of patients experience short-term postoperative voiding dysfunction. In order to provide convincing evidence that there may be a benefit to omitting plicating sutures, this study will be powered to detect a substantial difference in voiding dysfunction - from 50% of patients down to 25% of patients. Using a chi-square distribution and an alpha error of 0.05, the required sample size is 58 patients per group. (SAS 9.2)

Statistical Analysis Statistical analysis will be performed using SAS 9.2 for Windows™. Chi-square analysis will be used to evaluate categorical variables and T-Tests for continuous variables.

Data Management The data will be collected into a database. Statistical analysis will be conducted using SAS 9.2. All data will be kept confidential and protected.

Ethical Issues Written consent will be obtained from each participant. All data will be anonymous and will only be coded by a participant identification number.

An ethics proposal will be submitted to the Mount Sinai Hospital Research Ethics Board prior to beginning the recruitment. Patients with questions or concerns are free to contact the research assistant or a representative from the ethics board for clarification. The contact information will be noted in the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years, who will undergo surgery at the Mount Sinai Hospital that includes cystocele repair, will be eligible.

Exclusion Criteria:

* Patients will be excluded if the surgeon places anterior vaginal mesh or a mid-urethral sling, and/or if they had prior surgery for anterior vaginal wall prolapse and/or stress urinary incontinence.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Post operative voiding dysfunction | 24 hours post intervention
  The primary outcome variable will be the requirement for bladder catheterization beyond postoperative day 2

SECONDARY OUTCOMES:
Ureteric Obstruction | Intraoperative
  A secondary outcome will be intraoperative ureteric obstruction. All patients, regardless of study arm, will undergo intraoperative cystoscopy following intravenous administration of indigo carmine in order to identify this complication. If this complication does occur the suspected plicating suture(s) will removed, replaced more centrally, and cystoscopy repeated to ensure ureteric permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Lovatsis, MD, Principal Investigator — MOUNT SINAI HOSPITAL